CLINICAL TRIAL: NCT05416567
Title: Therapeutic Endovascular Embolization for Intracranial Meningioma
Brief Title: Embolization for Meningioma
Acronym: e-men
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 392999
Record Dates: First submitted 2022-05-09; First posted 2022-06-13 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Meningioma
Keywords: Brain neoplasms; Therapeutics
MeSH Terms: conditions — Meningioma; Brain Neoplasms

STUDY DESIGN:
Intervention Model Description: Historical controls from a regional brain tumor registry
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Endovascular embolization (Experimental)
  Interventions: Procedure: Endovascular embolization

INTERVENTIONS:
Procedure: Endovascular embolization — Therapeutic endovascular embolization in general anesthesia

SUMMARY:
The natural course for meningioma suggests that a majority will grow over time. Treatment is usually indicated in growing or symptomatic meningiomas. Surgery is usually primary treatment, but there is a significant risk of adverse effects. Stereotactic radiotherapy is most often reserved to treat relapses after surgery, and except for surgery and radiotherapy there are no other established treatment methods. Endovascular embolization may be used in selected cases as a preoperative adjunct to reduce intraoperative bleeding. There is a need for more treatment options in patients with meningioma, both in uncomplicated, asymptomatic cases and in more complex cases. The aim of this study is to assess radiological and clinical results of therapeutic endovascular embolization for meningioma

ELIGIBILITY:
Inclusion Criteria:

* Radiological diagnose of typical intracranial meningioma (homogenous contrast enhancement or dural attachment)
* Indication for treatment due to growth, symptoms or both
* Tumor location suggestive of vascular supply via middle meningeal artery branches
* Age 18 years or older
* Karnofsky performance status of 90 or better (able to carry on normal activity and work)

Exclusion Criteria:

* Informed consent not possible (e.g. language barriers, aphasia, cognitive impaired)
* Previously treated for meningioma
* Intraosseous growth
* Tumor related brain edema
* Neurofibromatosis type 2
* Systemic cancer
* Epilepsy
* Progressive neurodegenerative disorder (eg. MS, Parkinsons disease)
* History of psychiatric disorder
* Unfit for participation for any other reason judged by the physician including patients
* Contraindications to MRI
* Allergic to contrast agents
* Relative contraindications to endovascular treatment judged from CT angiography (tortoise carotid arteries, carotid stenosis, calcified aortic arch, anatomical vascular variants/anomalies suggesting increased risk with endovascular treatment)
* DSA (Digital subtraction angiography) from carotid artery suggesting that significant vascular supply is from other vessels than the MMA.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-10-10 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2037-08 (Estimated)

PRIMARY OUTCOMES:
Change in radiological tumor volume from baseline | At 1 year, 3 year and 5 year
  Volumetric segmentation of tumor volume

SECONDARY OUTCOMES:
Number of participants undergoing re-intervention for meningioma or treatment complications | 10 years
  Surgery or radiotherapy
Number of participants with epileptic seizures | 10 years
Number of participants with moderate or severe procedure related complications within 30 days | 30 days
  Landriel Ibanez classification (grade 3 or 4 complications)
Change in generic health-related quality of life from baseline | At 1 months and 6 months
  EuroQol-5D 3L (EQ-5D 3L)
Change in disease-specific quality of life from baseline | At 1 months and 6 months
  The European Organisation for Research and Treatment of Cancer (EORTC) QLQ-C30 questionnaire
Change in domain-specific quality of life from baseline | At 1 months and 6 months
  The European Organisation for Research and Treatment of Cancer (EORTC) QLQ-BN20 questionnaire
Change in neurological function | At 1 month
  National Institutes of Health Stroke Scale (NIHSS)
Number of participants with adverse events | 30 days
  Landriel Ibanez classification
Number of participants returning to work | At 1 months and 6 months
Loss of functional level from baseline | At 1 month and 6 months
  >10 points in Karnofsky performance status

CONTACTS AND LOCATIONS:
Overall Officials: Ole Solheim, PhD, Principal Investigator — St Olavs Hospital, Trondheim University Hospital, Trondheim, Norway
Locations (1):
- St Olavs Hospital, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: No